CLINICAL TRIAL: NCT05935280
Title: Human Cold Pain - a Single-group, Randomized, Placebo-controlled, Adaptive, Factorial Crossover Trial
Brief Title: Mechanism of Human Cold Pain Perception - Involvement of TRPA1, TRPM8, Nav1.7 and Nav1.8
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Stefan Heber, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EK Nr: 1164/2023
Record Dates: First submitted 2023-06-28; First posted 2023-07-07 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Pain
Keywords: Psychophysics; Human physiology; Cold perception; Transient receptor potential ion channels; Voltage-gated sodium channels; Sensory neuron
MeSH Terms: conditions — Pain | interventions — Cold Temperature; A 967079; PF-05089771

STUDY DESIGN:
Intervention Model Description: This study is a randomized, placebo-controlled, crossover trial. The factors determining the conditions varied within individuals are 'TRPM8 inhibitor', 'TRPA1 inhibitor', 'Nav1.7 inhibitor', 'Nav1.8 inhibitor' each with the levels 'inhibitor' or 'control'. The design allows estimating the effect size caused by each factor alone, as well as the fractional inhibition achieved when all four channels are blocked. In a separate condition, the hypothesized action of lidocaine against nerve conduction, thus including cold-induced activity, is intended as positive control.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Room temperature injection (Placebo Comparator): Pain induced by intradermal injection of fluid with room temperature.
  Interventions: Other: Room temperature
- Cold temperature injection 1 (Placebo Comparator): Pain induced by intradermal injection of increasingly cold fluid down to 3°C.
  Interventions: Other: Cold temperature
- Cold temperature injection with lidocain (Active Comparator): Pain induced by intradermal injection of increasingly cold fluid down to 3°C including lidocain (unspecific sodium channel blocker).
  Interventions: Other: Cold temperature; Drug: Lidocain
- Cold temperature injection 2 (Placebo Comparator): Pain induced by intradermal injection of increasingly cold fluid down to 3°C.
  Interventions: Other: Cold temperature
- Cold temperature injection with PF-05105679 (Experimental): Pain induced by intradermal injection of increasingly cold fluid down to 3°C including PF-05105679 (specific TRPM8 antagonist).
  Interventions: Other: Cold temperature; Drug: PF-05105679
- Cold temperature injection with A-967079 (Experimental): Pain induced by intradermal injection of increasingly cold fluid down to 3°C including A-967079 (specific TRPA1 antagonist).
  Interventions: Other: Cold temperature; Drug: A967079
- Cold temperature injection with PF-05089771 (Experimental): Pain induced by intradermal injection of increasingly cold fluid down to 3°C including PF-05089771 (specific Nav1.7 antagonist).
  Interventions: Other: Cold temperature; Drug: PF-05089771
- Cold temperature injection with PF-06305591 (Experimental): Pain induced by intradermal injection of increasingly cold fluid down to 3°C including PF-06305591 (specific Nav1.8 antagonist).
  Interventions: Other: Cold temperature; Drug: PF-06305591
- Cold temperature injection with PF-05105679, A-967079, PF-05089771, PF-06305591 (Experimental): Pain induced by intradermal injection of increasingly cold fluid down to 3°C including PF-05105679 (TRPM8)-, A-967079 (TRPA1)-, PF-05089771 (Nav1.7)-, PF-06305591 (Nav1.8)- antagonist.
  Interventions: Other: Cold temperature; Drug: PF-05105679; Drug: A967079; Drug: PF-05089771; Drug: PF-06305591

INTERVENTIONS:
Other: Room temperature — Room temperature injection
  Arms: Room temperature injection
Other: Cold temperature — Cold temperature injection
  Arms: Cold temperature injection 1; Cold temperature injection 2; Cold temperature injection with A-967079; Cold temperature injection with PF-05089771; Cold temperature injection with PF-05105679; Cold temperature injection with PF-05105679, A-967079, PF-05089771, PF-06305591; Cold temperature injection with PF-06305591; Cold temperature injection with lidocain
Drug: Lidocain — Unspecific sodium channel blocker
  Other Names: Unspecific sodium channel blocker
  Arms: Cold temperature injection with lidocain
Drug: PF-05105679 — Specific antagonist of the TRPM8 ion channel
  Other Names: Specific TRPM8 antagonist
  Arms: Cold temperature injection with PF-05105679; Cold temperature injection with PF-05105679, A-967079, PF-05089771, PF-06305591
Drug: A967079 — Specific antagonist of the TRPA1 ion channel
  Other Names: Specific TRPA1 antagonist
  Arms: Cold temperature injection with A-967079; Cold temperature injection with PF-05105679, A-967079, PF-05089771, PF-06305591
Drug: PF-05089771 — Specific antagonist of the Nav1.7 sodium channel
  Other Names: Specific Nav1.7 antagonist
  Arms: Cold temperature injection with PF-05089771; Cold temperature injection with PF-05105679, A-967079, PF-05089771, PF-06305591
Drug: PF-06305591 — Specific antagonist of the Nav1.8 sodium channel
  Other Names: Specific Nav1.8 antagonist
  Arms: Cold temperature injection with PF-05105679, A-967079, PF-05089771, PF-06305591; Cold temperature injection with PF-06305591

SUMMARY:
Animal studies suggest that the transient receptor potential ion channels TRPM8 and TRPA1 are cold sensors and that sodium channels Nav1.8 and Nav1.7 are essential for detecting pain induced by cold temperatures. This study aims to validate these findings in humans.

DETAILED DESCRIPTION:
It is essential for human survival to be able to perceive potentially harmful cold. The perception of slight cooling in animals depends on the ion channel TRPM8, but this may represent a largely separate mechanism from painful cold. In mice, TRPM8 and TRPA1 appear to be involved, but also the sodium channels Nav1.7 and Nav1.8, through their temperature-dependent function. These receptors might be redundant, so that failure of individual receptors only leads to no or only a partial reduction in the detection of cold.

Since results obtained in animals do not always translate to humans, the investigators want to clarify whether TRPM8, TRPA1, Nav1.7 and Nav1.8 are involved in the perception of cold pain in humans.

In order to induce cold pain experimentally, an increasingly cooled solution (down to 3°C) is injected into the skin, and the inhibitors for the mentioned targets are added individually and in combination.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Full legal capacity

To ensure an equal number of each sex in the study population, only volunteers of one sex will be included as soon as the number of subjects with the other sex has reached half of the calculated sample size.

Exclusion Criteria:

* Participant of another study, ongoing or within the last 4 weeks
* Medication intake (except contraception) or drug abuse
* Female subjects: Positive pregnancy test or breastfeeding
* Body temperature above 38°C, diagnostically verified
* Known allergic diseases, in particular asthmatic disorders and skin diseases
* Sensory deficit, skin disease or hematoma of unknown origin in physical examination of the test site

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
AUC Pain3°C | Through study completion, on average 90 minutes.
  The primary outcome variable is the area under the curve (AUC) of pain ratings over a limited duration of the infusion period, i.e. from 120-150 seconds (last 30 seconds of the cold stimulus).

SECONDARY OUTCOMES:
AUC Pain | Through study completion, on average 90 minutes.
  The secondary outcome variable is the area under the curve (AUC) of pain ratings over the full duration of the infusion period (full 150 seconds of the cold stimulus).

CONTACTS AND LOCATIONS:
Overall Officials: Michael JM Fischer, Study Chair — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
All raw data will be shared with other researches upon reasonable request.
Supporting Information: Study Protocol, Analytic Code
Time Frame: As soon as the study is published.
Access Criteria: Access will be granted to other researchers as well as clinicians.

REFERENCES:
- [Derived] Resch FJ, Heber S, Shahi F, Zauner M, Ciotu CI, Gleiss A, Sator S, Fischer MJM. Human cold pain: a randomized crossover trial. Pain. 2025 Jun 1;166(6):1406-1417. doi: 10.1097/j.pain.0000000000003503. Epub 2024 Dec 17. PMID 39693244